CLINICAL TRIAL: NCT07193979
Title: Relationship Between Diabetes and Periodontal Status and Dental Caries
Brief Title: Relationship Between Diabetes and Periodontitis
Status: Completed | Type: Observational
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Kübra Karaçam, assist. prof., Afyonkarahisar Health Sciences University
Other Study IDs: 2024/341
Record Dates: First submitted 2025-09-12; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Diabetes (DM); Periodontitis
MeSH Terms: conditions — Diabetes Mellitus; Periodontitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: HgA1c <7 diabetic patients
- Group 2: Diabetic patients with HgA1c 7≤ <8 in this range
- Group 3: HgA1c ≥8 diabetic patients

SUMMARY:
Diabetes mellitus, one of the major global health problems of the 21st century, is a chronic metabolic disease characterized by dysregulated nutrient metabolism resulting from defects in insulin secretion and action. Patients with diabetes mellitus are more likely to develop chronic periodontitis. A bidirectional relationship between diabetes mellitus and periodontitis has been demonstrated. Dental complications of diabetes mellitus include periodontitis and dental caries. Dental caries, resulting from tooth demineralization, are more prevalent in diabetic individuals than in non-diabetic individuals. For adults, HbA1c levels were defined as <7% ("good" control), HbA1c levels between 7% and 8% as "inadequate" control, and levels above 8% as "poor" control. In the study conducted by the investigators, patients diagnosed with type 2 diabetes mellitus and those diagnosed with periodontitis were grouped according to HbA1C levels, and the relationship between these levels and the stage/degree of periodontitis and the degree of caries was examined. Although studies on periodontal diseases and dental caries among adults with type 2 diabetes mellitus exist in the literature, no study has, as far as is known that classifies HbA1c levels in patients with controlled and uncontrolled diabetes diagnosed with periodontitis and explains the relationship between these groups and the stage/degree of periodontitis and the degree of caries.

DETAILED DESCRIPTION:
Mechanisms by which diabetes mellitus affects the periodontium have been reported, including altering host immune, inflammatory, and wound-healing responses, promoting the accumulation of advanced glycation end products, and inducing elevated levels of proinflammatory cytokines. Periodontitis is a common chronic infectious disease that can lead to the destruction of periodontal supporting tissues. Pathologically, a hyperactive inflammatory response contributes to the progression of these two diseases. Diabetes mellitus, in particular, increases the risk of periodontitis by activating immune and inflammatory responses in periodontal tissues. These active responses lead to increased cytokine secretion, increased oxidative damage, and impaired receptor-mediated signaling. All of these events accelerate the breakdown of periodontal connective tissue and alveolar bone resorption, thereby exacerbating periodontitis. Conversely, periodontitis can lead to deranged glycemic control in diabetic patients. Dental complications of diabetes mellitus include periodontitis and dental caries. Dental caries, resulting from tooth demineralization, is more prevalent in diabetic individuals than in non-diabetic individuals. The combination of carbohydrate intake and insulin deficiency leads to hyposalivation and higher salivary glucose levels, both of which contribute to an increased risk of dental caries. Factors that increase the risk of dental caries include decreased plaque microbial flora, decreased buffering and cleansing activities of saliva, decreased salivary flow rate, and decreased calcium levels. Glycemic control can be measured in various ways. For this study, researchers focused on glycated hemoglobin (HbA1c), which represents the average blood glucose levels over the previous 3 months. The study examined the relationship between the severity of periodontitis and the DMFT index according to HgA1C levels in diabetic patients. To our knowledge, no studies in the literature have classified HbA1c levels in patients with and without periodontitis, explaining the relationship between these groups and the stage/degree of periodontitis and the degree of caries. A standard periodontal examination was performed on the volunteers included in the study, and the gingival index (GI) (Loe & Silness, 1963 ), plaque index (PI) (Silness & Loe, 1964 ), probing depth (PD), bleeding on probing (BOP) (Ainamo & Bay, 1975 ), and clinical attachment level (CAL) were determined at six sites for each tooth except the third molars. The Decayed, Missing, and Filled Teeth (DMFT) index, declared by the World Health Organization, is an indicator of caries experience. During the intraoral examination, the total number of teeth and the status of teeth and fillings were recorded. Decayed teeth were examined visually and by radiographs. The numbers of decayed teeth (DT), missing teeth (MT), and filled teeth (FT) were recorded, and the DMFT index was calculated as the sum of DT+MT+FT.

ELIGIBILITY:
Inclusion Criteria:

Age between 20 and 65 years Diagnosed with Type 2 Diabetes Mellitus (T2DM) Diagnosed with periodontitis, according to established clinical criteria

Exclusion Criteria:

Diagnosis of Type 1 Diabetes Mellitus Diagnosis of gestational diabetes Presence of physical or mental disorders that may affect participation or evaluation Undergoing chemotherapy or radiotherapy Presence of any systemic disease other than diabetes mellitus Use of systemic antibiotics or other medications in the past 3 months Use of antiparkinsonian, antidepressant, or antipsychotic medications

Ages: 23 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study was conducted among individuals who applied to Afyonkarahisar Health Sciences University Faculty of Dentistry and volunteered to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Periodontal Index (PI) Score | One-time measurement at the beginning of the study
  PI will be used to assess periodontal health, scored according to WHO guidelines (Unit of Measure: Millimeters (mm))
Clinical Attachment Loss (CAL) | One-time measurement at the beginning of the study
  Clinical attachment loss will be measured at six sites per tooth using a periodontal probe (Unit of Measure: Millimeters (mm))
Probing Depth (PD) | One-time measurement at the beginning of the study
  Probing depth will be measured at six sites per tooth using a periodontal probe.(Millimeters (mm))
Total DMFT Index Score | One-time measurement at the beginning of the study
  The DMFT index will be calculated by summing the number of decayed (D), missing (M), and filled (F) teeth for each participant, as per WHO guidelines.

SECONDARY OUTCOMES:
Bleeding on Probing (BOP) | One-time measurement at the beginning of the study
  Bleeding on probing will be measured at six sites per tooth. The percentage of sites showing bleeding upon gentle probing will be recorded.
Gingival Index (GI) | One-time measurement at the beginning of the study
  Gingival inflammation will be assessed using the Löe and Silness Gingival Index, which scores the severity of gingivitis on a scale from 0 to 3.
Number of Decayed Teeth (D Component of DMFT Index) | One-time measurement at the beginning of the study
  The number of decayed teeth will be recorded according to WHO criteria.
Number of Missing Teeth (M Component of DMFT Index) | One-time measurement at the beginning of the study
  The number of missing teeth due to caries will be recorded based on clinical and anamnestic data.
Number of Filled Teeth (F Component of DMFT Index) | One-time measurement at the beginning of the study
  The number of teeth with permanent restorations due to dental caries will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Afyonkarahisar Health Sciences University Faculty of Dentistry, Afyonkarahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
In order to protect participant privacy and act in accordance with the ethics committee decision, individual participant data will not be shared.